CLINICAL TRIAL: NCT02647840
Title: The Effects of Voice Therapy Based on the Estill Voice Model: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 185519
Record Dates: First submitted 2015-12-22; First posted 2016-01-06 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2016-10

CONDITIONS: Functional Dysphonia
Keywords: dysphonia; voice therapy
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voice therapy (Other): All participants will receive voice therapy based on the Estill model. This is very similar to our usual intervention.
  Interventions: Behavioral: voice therapy

INTERVENTIONS:
Behavioral: voice therapy — voice therapy based on Estill Voice Model The study will provide primarily direct intervention, i.e. working directly on the voice with voice exercises based on the Estill model of voice. This will be structured and hierarchical. Participants will work through the content one-to-one with the voice specialist SLT at their level and pace, to suit their specific vocal needs, again reflecting current clinical practice. Participants may need fewer or more than four sessions to gain the required skills. Should patients need more than six session of voice therapy to recover their voice fully, final assessment for the study purposes will be taken at session 6, and voice therapy will continue as required.
  Other Names: Estill voice model

SUMMARY:
This study wants to investigate treatment for patients with common voice disorders where no surgical or medical treatment is needed. A voice disorder is when your voice is croaky, hoarse or when you lose it altogether. This can be a serious problem for people as it stops them from participating in their normal life (for example in their jobs, hobbies, family and wider social life).

This study will look at our most commonly used method of treatment for voice problems. This method is based on physical exercises which work on the muscles which produce the voice. This voice work was originally developed by Jo Estill, a singer and scientist, and is widely used in voice coaching. Though many Speech and Language Therapists (SLTs) provide voice therapy based on the Estill model, there is no clinical evidence to support its use.

The aim of this study is to test the design for a larger research study into the effects of voice therapy based on Estill model of voice. We want to find out if our tests work and are easy to use, and to check that the study methods are right and would work on a larger scale. It is a feasibility study, and therefore allows us to test whether this study can be done. Another important part of this study is to involve patients in developing research. We want to find out what patients think about the treatment they receive, and about taking part in a study.

The way this study will work is that patients who have agreed to take part will have between four and six voice therapy appointments, just like they would if they were not part of the study. Voice test results from before and after treatment will be compared and carefully studied. After patients taking part in the study have finished their treatment, they will be asked about their experience of voice therapy, and of being in the study. Much of what will be done as part of the study is identical to what is normally done in treatment, however we will look in detail at all the tests, and we need permission from participants to use their test results and include their comments.

It is important to learn more about voice therapy and to improve voice therapy for patients with this type of voice problem. By finding out more what patients think about the treatment we provide, what tests to use, and about how best to run a research trial, we will be able to plan further research and hopefully be successful at a next large research grant application.

DETAILED DESCRIPTION:
Aims and Objectives The overall aim of this study is to test the feasibility of a study into the effects of Estill based voice therapy for patients with functional dysphonia.

The objectives are:

To gather information that will help us design a larger study, specifically

* how many participants can we expect to recruit
* what is the rate of consent
* what is the rate of attrition
* how many therapy sessions do patients attend over what length of time (length episode of care & total therapy time in minutes) To test our outcome measures
* is using OperaVOX on iPad for clinical outcome measurement useful for clinician and participant; is it quick, easy to use, and reliable?
* what is the Standard Deviation (SD) for outcome measures so that we can estimate sample size for a further trial To describe therapy content in detail so that it can be replicated and meaningfully practised by participants
* what advice sheets/ therapy instructions do we give To investigate participant experience
* What is it like to have functional dysphonia
* What is it like to have voice therapy
* What is it like to take part in a study
* Does the overall design work smoothly for participants
* What worked well/ what could be better for participants Plan of investigation General research design This is a feasibility study using a mixed method research design. We will gain quantitative data from clinical voice assessments that will be analysed using descriptive statistics. We will also use qualitative research design when we use post-intervention focus groups to evaluate participants' experiences.

The study design does not control bias as it is not controlled and participants are not blinded to the intervention. We will therefore not be able to make a judgment as to whether Estill based voice therapy is effective in treating functional dysphonia in this study.

Study population The target population is adult patients referred into the SLT department by the Ear Nose Throat Consultant with a diagnosis of 'functional dysphonia', 'hyperfunctional dysphonia' or 'muscle tension dysphonia' and presenting with altered voice quality and essentially normal larynx on examination. Patients with a diagnosis of '(early) vocal nodules' and 'mild vocal oedema' may also be included as the underlying aetiology is inappropriate muscular tension and hyperfunction, and voice therapy the treatment of choice. Patients are aged 16 and above, and from Exeter, Mid and East Devon - the area normally served by the voice specialist service at the Royal Devon & Exeter Foundation NHS Trust.

We plan to include 20 patients, as this sample size will be adequate for making accurate estimations of recruitment and judgements about outcome measures (including SD).

Patients with voice problems that indicate the presence of muscle tension and diagnoses specified above are eligible to take part. Patients with hearing problems, cognitive difficulties such as memory loss, and significant co-morbidities such as uncontrolled reflux or previous radiotherapy for Head & Neck Cancer are excluded from the study, as these can limit expected progress. For the same reasons, patients with significant psychogenic issues underlying the voice problem will be excluded as they essentially have a diagnosis of psychogenic dysphonia. All patients not included in the study will be offered voice therapy as appropriate to their needs as usual.

Last year, 130 patients with functional dysphonia attended for voice therapy at the SLT department who would have been eligible to take part. It is estimated that it is feasible to recruit 20 participants over a six month period.

Potential participants will be identified on the basis of their referral letter from the ENT with diagnosis and presentation. When patients receive a standard letter inviting them to contact the SLT department for a voice therapy appointment, potentially eligible patients will receive an information leaflet about the study. On initial attendance at the SLT department, they will be given further information and a consent form to sign if they are happy to take part. It will be made clear that participants are free not to take part or to withdraw from the study at any time without it affecting their treatment in any way.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of muscle tension dysphonia or functional dysphonia

Exclusion Criteria:

* hearing problems, cognitive difficulties such as memory loss, and significant co-morbidities such as uncontrolled reflux or previous radiotherapy for Head & Neck Cancer; significant psychological issues underlying the voice problem

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03-28 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index 10 | at initial and final assessment, before after therapy (approx 3 month interval)
  Patient report questionnaire (Using OperavOx app)

SECONDARY OUTCOMES:
Qualitative feedback | after intervention, within 6 weeks of discharge
  Feedback form participants about the therapy and study given to independent researcher in small group interview after therapy

OTHER OUTCOMES:
Patient rating of their own therapy goal | at initial and final assessment, before and after therapy (approx 3 month interval)
  Participants define their own clinical goals and rate on 0-10 scale
Perceptual Voice Rating | at initial and final assessment, before and after therapy (approx 3 month interval)
  Perceptual rating of participant voice quality based on recorded samples, using GRBAS voice rating scale (Rough, Breathy, Strained parameter)
Maximum phonation time | at initial and final assessment, before and after therapy (approx 3 month interval)
  ability to sustain phonation (Using OperavOx app)
Acoustic voice analysis | at initial and final assessment, before and after therapy (approx 3 month interval)
  Acoustic analysis of voice sample: Jitter and Shimmer (Using OperavOx app)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm P Hilton, MD, Study Chair — Royal Devon and Exeter NHS Trust; Marianne E Bos-Clark, MSc, Principal Investigator — Royal Devon and Exter NHS Trust
Locations (1):
- Speech and Language Therapy Department, Royal Devon and Exeter NHS Foundation Trust (Wonford), Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No